CLINICAL TRIAL: NCT03480555
Title: Replacing Protein Via Enteral Nutrition in a Stepwise Approach in Critically Ill Patients: Feasibility Randomized Controlled Trial
Brief Title: Replacing Protein Via Enteral Nutrition in a Stepwise Approach in Critically Ill Patients
Acronym: Replenish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC17/252/R
Record Dates: First submitted 2018-02-22; First posted 2018-03-29 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Critical Illness; ARDS; Septic Shock; Multiple Trauma; Seizure Disorder; Hemorrhagic Shock
Keywords: Enteral nutrition, Intensive Care Units, caloric restriction, insulin, mortality, protein catabolism
MeSH Terms: conditions — Critical Illness; Shock, Septic; Multiple Trauma; Epilepsy; Shock, Hemorrhagic; Insulin Resistance | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Replenish Protein group (Active Comparator): Subjects randomized to this group will receive 2 g of protein/kg/day (acceptable range as 1.8 - 2.2 g of protein/kg/day) for day 6-14.
  Interventions: Dietary Supplement: Replenish Protein
- Standard Protein group (Other): Subjects randomized to this group will receive 0.8 - 1 g of protein/kg/day for day 6-14
  Interventions: Dietary Supplement: Standard protein

INTERVENTIONS:
Dietary Supplement: Replenish Protein — Subjects randomized to this group will receive 2 g of protein/kg/day (acceptable range as 1.8 - 2.2 g of protein/kg/day) for day 6-14.
  Other Names: Intervention group
  Arms: Replenish Protein group
Dietary Supplement: Standard protein — Subjects randomized to this group will receive 0.8 - 1 g of protein/kg/day for day 6-14
  Other Names: Control group
  Arms: Standard Protein group

SUMMARY:
In this study, we will explore the feasibility of a randomized controlled trial that will compare high protein dose from ICU day 6 to 14 with moderate protein intake.

DETAILED DESCRIPTION:
Patients will be recruited on day 1-2 of ICU admission. On day 5, patients will be randomized into one of the two intervention arms;

Replenish Protein group:

Patients randomized to this group will receive 2 g of protein/kg/day (acceptable range 1.8 - 2.2 g of protein/kg/day) for day 6-14.

Standard Protein group:

Patients randomized to this group will receive protein at 0.8 - 1.0 g of protein/kg/day for day 6-14

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years
2. Mechanically ventilated
3. Receiving enteral feeding via nasogastric/orogastric or duodenal or PEG or jejunostomy tubes and
4. Expected to stay ≥ 1 week in the ICU

Exclusion criteria

1. Lack of commitment to ongoing life support, which includes;

   * Terminal Illness (Malignancy or irreversible condition with 6 month mortality > 50%)
   * DNR order in the first 48 hours and brain death within 48 hours of admission) (Don't include the presence of a "Do Not Resuscitate" order alone, if there is a commitment to ongoing life support).
2. Patients not fed within 48 hours of admission
3. Patients on total parenteral nutrition (TPN)
4. Patients being fed orally
5. Chronic renal failure
6. Chronic liver disease
7. Renal replacement therapy
8. Pregnancy.
9. Kidney transplant
10. Post-liver transplant.
11. Post cardiac arrest.
12. Burn patients.
13. Prisoners

Screened patients will be screened again for eligibility at day 5, should be mechanically ventilated and expected to stay ≥ 3 days in the ICU. At this point, patients will be excluded if they meet the following;

1. New onset renal replacement therapy.
2. Acute Kidney Injury (serum creatinine > 3 times the preacute level or serum creatinine >350mmol/L with a recent increase of >44 mmols/L)
3. Significant liver impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Recruitment | 6 months
  Recruitment log
Retention rate | 14 days
  withdrawals
Achieved protein intake | 14 days
  Feeding data

CONTACTS AND LOCATIONS:
Overall Officials: Yaseen M Arabi, MD, Principal Investigator — King Abdulaziz Medical City-Ministry of National Guard
Locations (2):
- Saudi Arabia (2):
  - King Abdulaziz Medical city, Jeddah
  - King Abdulaziz Medical city, Riyadh

IPD SHARING:
Plan to Share IPD: No
Data will be shared with the other participating sites after the completion of the main study and upon the descretion of the study Principle investigator only

REFERENCES:
- [Result] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Result] Arabi YM, Aldawood AS, Solaiman O. Permissive Underfeeding or Standard Enteral Feeding in Critical Illness. N Engl J Med. 2015 Sep 17;373(12):1175-6. doi: 10.1056/NEJMc1509259. No abstract available. PMID 26376142
- [Result] Arabi YM, Casaer MP, Chapman M, Heyland DK, Ichai C, Marik PE, Martindale RG, McClave SA, Preiser JC, Reignier J, Rice TW, Van den Berghe G, van Zanten ARH, Weijs PJM. The intensive care medicine research agenda in nutrition and metabolism. Intensive Care Med. 2017 Sep;43(9):1239-1256. doi: 10.1007/s00134-017-4711-6. Epub 2017 Apr 3. PMID 28374096
- [Derived] Arabi YM, Al-Dorzi HM, Tamim H, Sadat M, Al-Hameed F, AlGhamdi A, Al Mekhlafi GA, Rasool G, Afesh L, Sakkijha MH, Alamrey NK, Malebari R, Alhutail RH, Al-Dawood A; Saudi Critical Care Trials Group. Replacing protein via enteral nutrition in a stepwise approach in critically ill patients: A pilot randomized controlled trial (REPLENISH pilot trial). Clin Nutr ESPEN. 2021 Aug;44:166-172. doi: 10.1016/j.clnesp.2021.05.008. Epub 2021 Jun 2. PMID 34330462